CLINICAL TRIAL: NCT04044352
Title: A Controlled Human Infection Study of Influenza A/Bethesda/MM2/H1N1 Virus (A/California/04/2009/H1N1-like) in Healthy Subjects to Assess the Effect of Pre-Existing Immunity on Symptomatic Influenza Virus Infection
Brief Title: H1N1v Virus Challenge Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-0010; HHSN272201300015I
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-12-29

CONDITIONS: Influenza
Keywords: A/Bethesda/MM2/H1N1 Virus; Challenge; Dose Escalation; Healthy Subjects; Influenza; Live virus
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1 (Experimental): 2 mL (approximately 5x10^6/mL tissue culture infective dose (TCID50)) of influenza A/Bethesda/MM2/H1N1challenge virus administered intranasally via a sprayer on Day 1. N=80.
  Interventions: Biological: Influenza A/Bethesda/MM2/H1N1 Challenge

INTERVENTIONS:
Biological: Influenza A/Bethesda/MM2/H1N1 Challenge — Reverse-genetics derived live A/California/04/2009/H1N1-like influenza virus passaged six times in Vero cells.

SUMMARY:
This is a study of a reverse-engineered, Good Manufacturing Practice (GMP) grade, antiviral-sensitive, influenza A/Bethesda/MM2/H1N1 virus (A/California/04/2009/H1N1-like) infection to assess the effect of pre-existing immunity on clinical and immunological responses. Up to 80 healthy adult subjects will undergo intranasal inoculation with A/Bethesda/MM2/H1N1 virus, and their clinical manifestations, viral shedding and immunological responses will be characterized. The Primary Objective for this study is to evaluate the association of symptomatic Reverse Transcription-Polymerase Chain Reaction (RT-PCR)-positive influenza virus infection post-challenge and pre-existing Hemagglutinin Inhibition Test (HAI) antibody titers.

DETAILED DESCRIPTION:
This is a study of a reverse-engineered, Good Manufacturing Practice (GMP) grade, antiviral-sensitive, influenza A/Bethesda/MM2/H1N1 virus (A/California/04/2009/H1N1-like) infection to assess the effect of pre-existing immunity on clinical and immunological responses. Up to 80 healthy adult subjects will undergo intranasal inoculation with A/Bethesda/MM2/H1N1 virus, and their clinical manifestations, viral shedding and immunological responses will be characterized. This proposed study will establish a H1N1 influenza virus controlled human infection (CHI) model at the National Institute of Allergy and Infectious Diseases (NIAID) Division of Microbiology and Infectious Diseases (DMID)-sponsored Vaccine and Treatment Evaluation Units (VTEU) clinical study sites. The model has been developed and used by NIAID Division of Intramural Research. The proposed study will expand US research capacity to perform influenza CHI studies to advance the understanding of influenza pathogenesis and novel vaccine research and development. The Primary Objective for this study is to evaluate the association of symptomatic Reverse Transcription-Polymerase Chain Reaction (RT-PCR)-positive influenza virus infection post-challenge and pre-existing Hemagglutinin Inhibition Test (HAI) antibody titers. The Secondary Objectives for this study are: 1) To describe viral recovery by quantitative RT-PCR from study subjects at baseline and post-challenge; 2) To describe serum HAI and MN antibody responses post-challenge in healthy subjects by infection status; 3) To evaluate the association of asymptomatic RT-PCR-positive influenza virus infection (viral shedding) post-challenge and pre-existing HAI antibody titers; 4) To evaluate the association of symptomatic RT-PCR-negative status post-challenge and pre-existing HAI antibody titers; 5) To determine the frequency of serious adverse events (SAE) post-challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedure.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Agree to remain an inpatient for at least seven days after challenge, and until they have no virus shedding,* determined by qualitative RT-PCR for a minimum of two consecutive days post-challenge.

   * For a minimum of seven days post-challenge (Study Day 8).
4. Healthy* males and non-pregnant, non-breastfeeding females**, aged >/= 18 and </=49 years of age, inclusive, at enrollment.

   *Good health is defined in inclusion criteria 10.
   * Females subjects of childbearing potential must agree to have a serum pregnancy test at screening, a urine pregnancy test before Chest X-Ray (CXR) performed (if more than 7 days have passed between CXR and serum pregnancy test), and a urine pregnancy test upon admission to the inpatient unit prior to CHI, and results must be negative.
5. Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least 1 acceptable primary form of contraception***,****.

   These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).

   *Not of child bearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure(R) placement with history of documented radiological confirmation test at least 90 days after the procedure).

   **True abstinence is 100% of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

   ***Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for180 days or more prior to the subject receiving the influenza challenge virus, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products.

   ****Must use at least one acceptable primary form of contraception for at least 30 days prior to admission and at least one acceptable primary form of contraception during the remainder of the study.
6. Non-habitual smoker* of tobacco, e-cigarettes or marijuana.

   *Non-habitual smokers are those who smoke no more than four cigarettes, other tobacco products, e-cigarettes or marijuana in a week for more than three months and agree not to smoke cigarettes, other tobacco products, e-cigarettes and/or marijuana products during participation in the study.
7. No self-reported or known history of alcoholism or drug use within the last 30 days and agrees to abstain from alcohol and drugs* for at least one week before admission and throughout the inpatient period.

   *Including forms of marijuana not included in criterion 6.
8. Negative drug urine toxicology result on screening (i.e., amphetamines, cocaine, and opiates) and on admission to the challenge unit (i.e., amphetamines, cocaine, opiates, and cannabinoids).
9. Agree not to use the listed* prescription or over-the-counter medications within 7 days prior to inpatient stay and through inpatient stay, unless approved by the investigator.

   *Oseltamivir, zanamivir, peramivir, baloxavir marboxil, amantadine (generic) and rimantadine (Flumadine and generic), aspirin, intranasal steroids, decongestants, antihistamines, and other non-steroidal anti-inflammatory drugs (NSAIDs).
10. In good health* and not have clinically significant medical, psychiatric, chronic or intermittent health conditions including those listed in the Subject Exclusion Criteria.

    *Good health, as determined by medical history, medication use and physical examination to evaluate ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would not affect the assessment of the safety of subjects or the immunogenicity of challenge. These medical diagnoses or conditions should be stable for the last 90 days (no hospitalizations, emergency room (ER) or urgent care for condition (excluding musculoskeletal conditions) and not listed in the Subject Exclusion Criteria. Subjects may be on medications only if the condition or disease is stable and not deteriorating, if the medical intervention (such as device or medication) was not available during the maximal inpatient period of time, medications are not listed in the Subject Exclusion Criteria and pose no additional risk to subject safety or assessment of adverse events. This also includes no change in prescription medication, dose or frequency as a result of new symptoms or deterioration of the medical diagnosis or condition in the 90 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome (e.g., lowering of the dosage or frequency), as determined by the site principal investigator (PI) or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572, will not be considered a deviation of this inclusion criterion.
11. Does not have an ongoing symptomatic condition* for which subject has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan.

    *e.g., ongoing fatigue without a diagnosis for symptom.
12. Vital signs as follows: pulse is 47 to 99 beats per minute, inclusive; systolic blood pressure is 85 to 139 mmHg, inclusive; diastolic blood pressure is 55 to 89 mmHg, inclusive; SpO2 >95%; RR<18; oral temperature is less than 100.0 Degrees Fahrenheit.
13. Eligibility laboratory values (White Blood Cell (WBC), Absolute Lymphocyte Count, Hemoglobin (Hgb), Platelets (PLTs), Alanine Transaminase (ALT) and Creatinine (Cr)) are within acceptable parameters.
14. Body mass index (BMI) >18.5 and <35 kg/m^2 at screening.
15. Other screening tests (ECG and CXR) are within normal reference range or not deemed clinically significant by the PI or appropriate sub-investigator*.

    *Designated clinician licensed to make medical diagnoses and listed on the Form FDA 1572.
16. Negative test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) at screening blood draw.
17. Negative respiratory virus panel by BIOFIRE(R) FILMARRAY(R) respiratory panel by bioMérieux or by Luminex xTAG (R) on Day (-2), and Day (-1).

Exclusion Criteria:

1. Female subject who has a positive pregnancy test on screening or admission, is breastfeeding or planning to become pregnant from 30 days prior to challenge through the end of the study.
2. Presence of self-reported or medically documented significant medical or psychiatric condition(s)*.

   *Significant medical or psychiatric conditions include but are not limited to:
   * Respiratory disease (e.g., chronic obstructive pulmonary disease (COPD), asthma) requiring daily medications (Asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics) currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years
   * Presence of any febrile illness or symptoms suggestive of a respiratory infection within two weeks prior to Controlled Human Infection (CHI).
   * Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
   * Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures, encephalopathy, focal neurologic deficits, Guillain-Barre syndrome, encephalomyelitis or transverse myelitis).
   * Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell carcinoma of the skin, which is allowed.
   * An autoimmune disease.
   * An immunodeficiency of any cause.
   * A history of diabetes.
3. Presence of immunosuppression or any medications that may be associated with impaired immune responsiveness*.

   *Including, but not limited to, corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids or other similar or toxic drugs during the preceding 12-month period prior to screening. Low dose topical and intranasal steroid preparations used for a discrete period of time are permitted.
4. Known allergy or intolerance to treatments for influenza (including but not limited to oseltamivir, baloxavir marboxil, acetaminophen).
5. Known allergy to two or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
6. Known allergy to excipients in the challenge virus inoculum.
7. Receipt or planned receipt of any investigational drug/investigational vaccine/licensed vaccine within 30 days prior to the date of CHI.
8. Prior enrollment in any influenza virus challenge study.
9. Currently enrolled in any investigational study or intends to enroll in such a study within the ensuing study period.
10. Receipt of any influenza vaccine six months prior to challenge or plans to receive influenza vaccine within 60 days post-challenge.
11. History of a previous severe allergic reaction of any kind with generalized urticaria, angioedema, or anaphylaxis.
12. Receipt of blood or blood products during the six months prior to the planned date of challenge.
13. History of blood donation during the two months prior to the planned date of challenge and or plans to donate blood for the duration of the study.
14. Any condition, to include medical and psychiatric conditions, that in the opinion of the Investigator, might interfere with the safety of the subject and/or study objectives.
15. Known close contact with anyone known to have influenza 7 days prior to challenge.
16. Acute medical condition with new prescription medication use in the last 30 days.
17. Significant abnormality altering the anatomy of the nose/nasopharynx* clinically significant nasal deviation, or nasal/sinus surgery within 180 days prior to challenge.

    *Including significant nasal polyps.
18. History in the last five years of chronic or frequent intermittent sinusitis.
19. Recent history (180 days) of epistaxis or anatomic or neurologic abnormality impairing the gag reflex or contributing to aspiration.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Maryland Baltimore - School of Medicine - Medicine, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio

REFERENCES:
- [Derived] Ortiz JR, Bernstein DI, Hoft DF, Woods CW, McClain MT, Frey SE, Brady RC, Bryant C, Wegel A, Frenck RW, Walter EB, Abate G, Williams SR, Atmar RL, Keitel WA, Rouphael N, Memoli MJ, Makhene MK, Roberts PC, Neuzil KM. A Multicenter, Controlled Human Infection Study of Influenza A(H1N1)pdm09 in Healthy Adults. J Infect Dis. 2023 Aug 11;228(3):287-298. doi: 10.1093/infdis/jiad021. PMID 36702771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults, male and female, between the ages of 18 and 49, who are non-habitual smokers without medical conditions at high risk for severe complications of influenza virus infection were enrolled. Participants were enrolled between 22OCT2019 and 05DEC2019.
Groups:
- Study Group: Participants will receive 2 mL (approximately 5x10^6/mL tissue culture infective dose (TCID50)) of influenza A/Bethesda/MM2/H1N1 challenge virus administered intranasally via a sprayer on Day 1.
Period: Overall Study
Arm/Group | Study Group
Started | 76
Completed | 65
Not Completed | 11
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Study Group: Participants will receive 2 mL (approximately 5x10^6/mL tissue culture infective dose (TCID50)) of influenza A/Bethesda/MM2/H1N1challenge virus administered intranasally via a sprayer on Day 1.
Arm/Group | Study Group
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 34
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 76
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Saint Louis University | 17
  United States: Cincinnati Children's Hospital | 24
  United States: University of Maryland | 20
  United States: Duke University | 15
Receipt of Prior Seasonal Influenza Vaccination (2018-2019) [Count of Participants; unit: Participants]
  Yes | 9
  No | 67
Receipt of Prior Non-Seasonal Influenza Vaccination (2018-2019) [Count of Participants; unit: Participants]
  Yes | 3
  No | 73
Baseline Seroprotection (Hemagglutination Inhibition) [Count of Participants; unit: Participants]
  Low < 1:40 | 39
  High >= 1:40 | 37
Baseline Seroprotection (Microneutralization) [Count of Participants; unit: Participants]
  Low < 1:40 | 23
  High >= 1:40 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Healthy Participants Reporting Mild-to-Moderate Influenza Disease (MMID) by Baseline A/Bethesda/MM2/H1N1 Hemagglutination Inhibition (HAI) Antibody Seroprotection Status (Titer >/= 1:40 vs. Titer < 1:40)
Description: Blood samples were collected pre-challenge (Day -2) for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). MMID is a composite endpoint determined by the presence of viral shedding (detected by any approved positive RT-PCR test from a NP swab), accompanied by at least one the following symptoms occurring any time from Day 2 through Day 8; body aches or pain, chest tightness, chills, conjunctivitis, nasal congestion, sinus congestion, coryza, decreased appetite, diarrhea, dry cough, dyspnea, fatigue, fever, headache, lymphopenia, nausea, a 3% or more decrease in oxygen saturation from baseline, productive cough, rhinorrhea, sore throat, and sweats. The percentage of participants that developed MMID was calculated within each pre-challenge seroprotection status group.
Time Frame: Day 2 through Day 8
Population: All participants who received the study challenge, had a baseline sample for immunogenicity, and were followed for the entire duration of the study challenge period, or at least until MMID was observed.
Measure: Number; unit: percentage of participants
Groups:
- Study Group: 2 mL (approximately 5x10^6/mL tissue culture infective dose (TCID50)) of influenza A/Bethesda/MM2/H1N1 challenge virus administered intranasally via a sprayer on Day 1.
Arm/Group | Study Group
Number analyzed (Participants) | 76
percentage of participants
  Baseline Seroprotection Status Low < 1:40 : MMID: number analyzed (Participants) | 39
  Baseline Seroprotection Status Low < 1:40 : MMID | 77
  Baseline Seroprotection Status Low < 1:40 : No MMID: number analyzed (Participants) | 39
  Baseline Seroprotection Status Low < 1:40 : No MMID | 23
  Baseline Seroprotection Status High > = 1:40 : MMID: number analyzed (Participants) | 37
  Baseline Seroprotection Status High > = 1:40 : MMID | 65
  Baseline Seroprotection Status High > = 1:40 : No MMID: number analyzed (Participants) | 37
  Baseline Seroprotection Status High > = 1:40 : No MMID | 35

2. Primary Outcome: Association Between Clinical or Laboratory Manifestation of MMID and A/Bethesda/MM2/H1N1 HAI Antibodies in Serum at Baseline
Description: Blood samples were collected pre-challenge (Day -2) for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results. MMID is a composite endpoint determined by the presence of viral shedding (detected by any approved positive RT-PCR test from a NP swab), accompanied by at least one the following symptoms occurring any time from Day 2 through Day 8; body aches or pain, chest tightness, chills, conjunctivitis, nasal congestion, sinus congestion, coryza, decreased appetite, diarrhea, dry cough, dyspnea, fatigue, fever, headache, lymphopenia, nausea, a 3% or more decrease in oxygen saturation from baseline, productive cough, rhinorrhea, sore throat, and sweats. The relationship between the level of pre-challenge HAI titer and the likelihood of developing MMID during the study challenge period (Day 2 to Day 8) was assessed via logistic regression.
Time Frame: Day 2 to Day 8
Population: as for outcome 1
Measure: Number; unit: Odds Ratio
Groups:
- Study Group: 2 mL (approximately 5x10^6/mL tissue culture infective dose (TCID50)) of influenza A/Bethesda/MM2/H1N1challenge virus administered intranasally via a sprayer on Day 1.
Arm/Group | Study Group
Number analyzed (Participants) | 76
Odds Ratio | 0.81
Statistical Analysis 1: Comparison: Study Group; Pre-challenge (baseline) HAI geometric mean titer was log-2 transformed and treated as a continuous variable in the model; Test type: Other — Likelihood ratio test was the statistical test; p = 0.126, Wald Chi-Square; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.62 to 1.06] — A two-fold increase in HAI pre-challenge titer (i.e. one unit increase in log-2 titer) corresponds to a 19% decrease in the odds of developing MMID during the study challenge period (Day 2 through Day 8)

3. Secondary Outcome: Geometric Mean Titer (GMT) of HAI Antibody in Serum at Baseline by Infection Status
Description: Blood samples were collected pre-challenge (Day -2) and post-challenge on Days 8, 29 and 61 for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results. The geometric mean across samples was calculated within each study day and by infection status as observed over the study challenge period (Day 2 to Day 8); RT-PCR Negative (never positive), RT-PCR Positive Asymptomatic (participants with at least one positive PCR result but no symptoms reported), at least once RT-PCR Positive Symptomatic (or MMID).
Time Frame: Day -2
Population: All participants who received the study challenge, had an available immunogenicity sample for the given study day, and were followed for the entire duration of the study challenge period, or at least until MMID was observed.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 76
titer
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 54
  RT-PCR Positive Symptomatic | 36.8 [26.1 to 52.0]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 8
  RT-PCR Positive Asymptomatic | 20.0 [6.9 to 58.0]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 117.9 [61.3 to 227.0]

4. Secondary Outcome: GMT of HAI Antibody in Serum at Day 8 by Infection Status
Description: as for outcome 3
Time Frame: Day 8
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 75
titer
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 53
  RT-PCR Positive Symptomatic | 46.1 [33.2 to 64.0]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 8
  RT-PCR Positive Asymptomatic | 23.7 [8.9 to 63.1]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 122.5 [66.9 to 224.6]

5. Secondary Outcome: GMT of HAI Antibody in Serum at Day 29 by Infection Status
Description: as for outcome 3
Time Frame: Day 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 67
titer
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 46
  RT-PCR Positive Symptomatic | 87.4 [65.7 to 116.2]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 7
  RT-PCR Positive Asymptomatic | 63.9 [29.2 to 139.9]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 126.6 [72.3 to 221.9]

6. Secondary Outcome: GMT of HAI Antibody in Serum at Day 61 by Infection Status
Description: as for outcome 3
Time Frame: Day 61
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 62
titer
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 43
  RT-PCR Positive Symptomatic | 78.0 [55.5 to 109.7]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 6
  RT-PCR Positive Asymptomatic | 71.3 [33.6 to 151.1]
  RT-PCR Negative: number analyzed (Participants) | 13
  RT-PCR Negative | 123.1 [63.9 to 237.3]

7. Secondary Outcome: Percentage of Healthy Participants Achieving HAI Seroconversion From Baseline in Serum at Day 8 by Infection Status
Description: Blood samples were collected pre-challenge (Day -2) and post-challenge on Days 8, 29 and 61 for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. Seroconversion was defined as a pre-challenge titer 1:10 or greater and a minimum 4-fold rise in post-challenge antibody titer. The percentage of participants achieving seroconversion was calculated within each post-challenge study day and by infection status as observed over the study challenge period (Day 2 to Day 8); RT-PCR Negative (never positive), RT-PCR Positive Asymptomatic (participants with at least one positive PCR result but no symptoms reported), at least once RT-PCR Positive Symptomatic (or MMID).
Time Frame: Day 8
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 75
percentage of participants
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 53
  RT-PCR Positive Symptomatic | 3.8 [0.5 to 13]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 8
  RT-PCR Positive Asymptomatic | 0 [0 to 36.9]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 0 [0 to 23.2]

8. Secondary Outcome: Percentage of Healthy Participants Achieving HAI Seroconversion in Serum From Baseline at Day 29 by Infection Status
Description: as for outcome 7
Time Frame: Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 67
percentage of participants
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 46
  RT-PCR Positive Symptomatic | 28.3 [16 to 43.5]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 7
  RT-PCR Positive Asymptomatic | 28.6 [3.7 to 71]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 0 [0 to 23.2]

9. Secondary Outcome: Percentage of Healthy Participants Achieving HAI Seroconversion in Serum From Baseline at Day 61 by Infection Status
Description: as for outcome 7
Time Frame: Day 61
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 62
percentage of participants
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 43
  RT-PCR Positive Symptomatic | 18.6 [8.4 to 33.4]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 6
  RT-PCR Positive Asymptomatic | 33.3 [4.3 to 77.7]
  RT-PCR Negative: number analyzed (Participants) | 13
  RT-PCR Negative | 0 [0 to 24.7]

10. Secondary Outcome: GMT of Microneutralization (MN) Antibody in Serum at Baseline by Infection Status
Description: Blood samples were collected pre-challenge (Day -2) and post-challenge on Days 8, 29 and 61 for the MN assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results. The geometric mean across samples was calculated within each study day and by infection status as observed over the study challenge period (Day 2 to Day 8); RT-PCR Negative (never positive), RT-PCR Positive Asymptomatic (participants with at least one positive PCR result but no symptoms reported), at least once RT-PCR Positive Symptomatic (or MMID).
Time Frame: Day -2
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 76
titer
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 54
  RT-PCR Positive Symptomatic | 62.9 [43.1 to 91.9]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 8
  RT-PCR Positive Asymptomatic | 44.3 [13.8 to 142.6]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 276.7 [124.8 to 613.1]

11. Secondary Outcome: GMT of MN Antibody in Serum at Day 8 by Infection Status
Description: as for outcome 10
Time Frame: Day 8
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 75
titer
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 53
  RT-PCR Positive Symptomatic | 87.7 [61.7 to 124.6]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 8
  RT-PCR Positive Asymptomatic | 52.4 [16.6 to 165.5]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 250.6 [112.8 to 556.9]

12. Secondary Outcome: GMT of MN Antibody in Serum at Day 29 by Infection Status
Description: as for outcome 10
Time Frame: Day 29
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 67
titer
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 46
  RT-PCR Positive Symptomatic | 159.5 [115.7 to 220.1]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 7
  RT-PCR Positive Asymptomatic | 103.1 [41.5 to 255.9]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 320.0 [157.9 to 648.5]

13. Secondary Outcome: GMT of MN Antibody in Serum at Day 61 by Infection Status
Description: as for outcome 10
Time Frame: Day 61
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group
Number analyzed (Participants) | 62
titer
  RT-PCR Positive Symptomatic (MMID-1): number analyzed (Participants) | 43
  RT-PCR Positive Symptomatic (MMID-1) | 151.8 [108.7 to 211.9]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 6
  RT-PCR Positive Asymptomatic | 107.2 [30.4 to 377.8]
  RT-PCR Negative: number analyzed (Participants) | 13
  RT-PCR Negative | 287.6 [134.9 to 613.2]

14. Secondary Outcome: Percentage of Healthy Participants Achieving MN Seroconversion From Baseline in Serum at Day 8 by Infection Status
Description: Blood samples were collected pre-challenge (Day -2) and post-challenge on Days 8, 29 and 61 for the MN assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. Seroconversion was defined as a pre-challenge titer 1:10 or greater and a minimum 4-fold rise in post-challenge antibody titer. The percentage of participants achieving seroconversion was calculated within each post-challenge study day and by infection status as observed over the study challenge period (Day 2 to Day 8); RT-PCR Negative (never positive), RT-PCR Positive Asymptomatic (participants with at least one positive PCR result but no symptoms reported), at least once RT-PCR Positive Symptomatic (or MMID).
Time Frame: Day 8
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 75
percentage of participants
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 53
  RT-PCR Positive Symptomatic | 7.5 [2.1 to 18.2]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 8
  RT-PCR Positive Asymptomatic | 0 [0 to 36.9]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 0 [0 to 23.2]

15. Secondary Outcome: Percentage of Healthy Participants Achieving MN Seroconversion From Baseline in Serum at Day 29 by Infection Status
Description: as for outcome 14
Time Frame: Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 67
percentage of participants
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 46
  RT-PCR Positive Symptomatic | 26.1 [14.3 to 41.1]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 7
  RT-PCR Positive Asymptomatic | 28.6 [3.7 to 71]
  RT-PCR Negative: number analyzed (Participants) | 14
  RT-PCR Negative | 0 [0 to 23.2]

16. Secondary Outcome: Percentage of Healthy Participants Achieving MN Seroconversion From Baseline in Serum at Day 61 by Infection Status
Description: as for outcome 14
Time Frame: Day 61
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 62
percentage of participants
  RT-PCR Positive Symptomatic: number analyzed (Participants) | 43
  RT-PCR Positive Symptomatic | 18.6 [8.4 to 33.4]
  RT-PCR Positive Asymptomatic: number analyzed (Participants) | 6
  RT-PCR Positive Asymptomatic | 50 [11.8 to 88.2]
  RT-PCR Negative: number analyzed (Participants) | 13
  RT-PCR Negative | 0 [0 to 24.7]

17. Secondary Outcome: Duration of Viral Shedding in Nasopharyngeal (NP) Swab by Baseline HAI Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). Duration of viral shedding (detected by any approved positive RT-PCR test from NP swab) was calculated from the day of the initial positive PCR result to the day of the last positive PCR result prior to discharge from the challenge unit facility, regardless of intermittent negative PCR results. The mean duration of viral shedding was calculated among participants with detected virus within each pre-challenge HAI seroprotection status group.
Time Frame: Day 2 through Day 15
Population: All participants who received the study challenge, had a baseline sample for immunogenicity, and were followed for the entire duration of the study challenge period.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Study Group
Number analyzed (Participants) | 61
days
  Low < 1:40: number analyzed (Participants) | 35
  Low < 1:40 | 3.8 [2.9 to 4.7]
  High >= 1:40: number analyzed (Participants) | 26
  High >= 1:40 | 2.3 [1.6 to 3.0]

18. Secondary Outcome: Duration of Viral Shedding in NP Swab by Baseline MN Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the MN assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). Duration of viral shedding (detected by any approved positive RT-PCR test from NP swab) was calculated from the day of the initial positive PCR result to the day of the last positive PCR result prior to discharge from the challenge unit facility, regardless of intermittent negative PCR results. The mean duration of viral shedding was calculated among participants with detected virus within each pre-challenge MN seroprotection status group.
Time Frame: Day 2 to Day 15
Population: as for outcome 17
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Study Group
Number analyzed (Participants) | 75
Days
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 3.9 [2.6 to 5.2]
  High >= 1:40: number analyzed (Participants) | 52
  High >= 1:40 | 2.7 [2.1 to 3.3]

19. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 2 by Baseline HAI Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated for available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). The number of participants with viral shedding (detected by any approved positive RT-PCR test from a NP swab) was calculated for each study day post-challenge (Day 2 to Day 8) and at any time during the entire challenge period within each pre-challenge seroprotection status group.
Time Frame: Day 2
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 35
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 25

20. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 3 by Baseline HAI Seroprotection Status
Description: as for outcome 19
Time Frame: Day 3
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 27
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 11

21. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 4 by Baseline HAI Seroprotection Status
Description: as for outcome 19
Time Frame: Day 4
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 18
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 7

22. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 5 by Baseline HAI Seroprotection Status
Description: as for outcome 19
Time Frame: Day 5
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 15
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 0

23. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 6 by Baseline HAI Seroprotection Status
Description: as for outcome 19
Time Frame: Day 6
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 12
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 3

24. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 7 by Baseline HAI Seroprotection Status
Description: as for outcome 19
Time Frame: Day 7
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 9
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 1

25. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 8 by Baseline HAI Seroprotection Status
Description: as for outcome 19
Time Frame: Day 8
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 75
Participants
  Low < 1:40: number analyzed (Participants) | 38
  Low < 1:40 | 5
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 1

26. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab Anytime Post-challenge by Baseline HAI Seroprotection Status
Description: as for outcome 19
Time Frame: Day 2 to Day 8
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 36
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 26

27. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 2 by Baseline MN Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the MN assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated for available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). The number of participants with viral shedding (detected by any approved positive RT-PCR test from a NP swab) was calculated for each study day post-challenge (Day 2 to Day 8) and at any time during the entire challenge period within each pre-challenge seroprotection status group.
Time Frame: Day 2
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 21
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 39

28. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 3 by Baseline MN Seroprotection Status
Description: as for outcome 27
Time Frame: Day 3
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 16
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 22

29. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 4 by Baseline MN Seroprotection Status
Description: as for outcome 27
Time Frame: Day 4
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 10
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 15

30. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 5 by Baseline MN Seroprotection Status
Description: as for outcome 27
Time Frame: Day 5
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 9
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 6

31. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 6 by Baseline MN Seroprotection Status
Description: as for outcome 27
Time Frame: Day 6
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 8
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 7

32. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 7 by Baseline MN Seroprotection Status
Description: as for outcome 27
Time Frame: Day 7
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 6
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 4

33. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab at Day 8 by Baseline MN Seroprotection Status
Description: as for outcome 27
Time Frame: Day 8
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 75
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 5
  High >= 1:40: number analyzed (Participants) | 52
  High >= 1:40 | 1

34. Secondary Outcome: Number of Participants With Viral Shedding in NP Swab Anytime Post-challenge by Baseline MN Seroprotection Status
Description: as for outcome 19
Time Frame: Day 2 through Day 8
Population: All participants who received the study challenge with available results.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 22
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 40

35. Secondary Outcome: Time Until Detectable Viral Shedding in NP Swab by Baseline HAI Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). Time until viral shedding (detected by any approved positive RT-PCR test from a NP swab) was calculated as the initial day of viral shedding post-challenge for each participant. Median time to viral shedding was calculated within each pre-challenge seroprotection status group via the Kaplan-Meier estimator.
Time Frame: Day 2 through Day 8
Population: All participants who received the study challenge, had a baseline sample for immunogenicity, and were followed for the entire duration of the study challenge period, or at least until viral shedding was observed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Study Group
Number analyzed (Participants) | 76
Days
  Low < 1:40: number analyzed (Participants) | 39
  Low < 1:40 | 2.0 [NA to NA] — Not calculable due to insufficient variability
  High >= 1:40: number analyzed (Participants) | 37
  High >= 1:40 | 2.0 [NA to NA] — Not calculable due to insufficient variability
  All Subjects | 2.0 [NA to NA] — Not calculable due to insufficient variability

36. Secondary Outcome: Time Until Detectable Viral Shedding in NP Swab by Baseline MN Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the MN assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). Time until viral shedding (detected by any approved positive RT-PCR test from a NP swab) was calculated as the initial day of viral shedding post-challenge for each participant. Median time to viral shedding was calculated within each pre-challenge seroprotection status group via the Kaplan-Meier estimator.
Time Frame: Day 2 through Day 8
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Study Group
Number analyzed (Participants) | 76
Days
  Low < 1:40: number analyzed (Participants) | 23
  Low < 1:40 | 2.0 [NA to NA] — Not calculable due to insufficient variability
  High >= 1:40: number analyzed (Participants) | 53
  High >= 1:40 | 2.0 [NA to NA] — Not calculable due to insufficient variability

37. Secondary Outcome: Magnitude of Viral Shedding in NP Swab by Baseline HAI Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). The quantity of viral load copies/mL from NP swab was measured via quantitative RT-PCR result for each post-challenge study day. The mean of each sample's quantitative PCR replicate results was calculated from available results. Total viral shedding, as observed until study discharge, was calculated as the area under the curve (AUC), then log-10 transformed. Peak viral shedding was calculated as the maximum viral load copies/mL observed until study discharge, then log-10 transformed. The mean and median of the log-10 AUC and the mean and median of the log-10 peak viral load were both calculated within each pre-challenge seroprotection status group.
Time Frame: Day 2 through Day 15
Population: All participants who received the study challenge, had a baseline sample for immunogenicity, were followed for the entire duration of the study challenge period,.
Measure: Mean (Full Range); unit: log-10 copies/mL
Arm/Group | Study Group
Number analyzed (Participants) | 75
log-10 copies/mL
  Peak viral load - Low < 1:40: number analyzed (Participants) | 38
  Peak viral load - Low < 1:40 | 4.7 [-1.5 to 14.8]
  Peak viral load - High >= 1:40: number analyzed (Participants) | 37
  Peak viral load - High >= 1:40 | 2.1 [-1.2 to 11.6]
  AUC - Low < 1:40: number analyzed (Participants) | 38
  AUC - Low < 1:40 | 4.7 [-2.2 to 14.8]
  AUC - High >= 1:40: number analyzed (Participants) | 37
  AUC - High >= 1:40 | 1.8 [-1.7 to 11.6]

38. Secondary Outcome: Magnitude of Viral Shedding in NP Swab by Baseline MN Seroprotection Status
Description: Blood samples were collected pre-challenge (Day -2) for the MN assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). The quantity of viral load copies/mL from NP swab was measured via quantitative RT-PCR result for each post-challenge study day. The mean of each sample's quantitative PCR replicate results was calculated from available results. Total viral shedding, as observed until study discharge, was calculated as the area under the curve (AUC), then log-10 transformed. Peak viral shedding was calculated as the maximum viral load copies/mL observed until study discharge, then log-10 transformed. The mean and median of the log-10 AUC and the mean and median of the log-10 peak viral load were both calculated within each pre-challenge seroprotection status group.
Time Frame: Day 2 through Day 15
Population: as for outcome 17
Measure: Mean (Full Range); unit: log-10 copies/mL
Arm/Group | Study Group
Number analyzed (Participants) | 75
log-10 copies/mL
  Peak viral load - Low < 1:40: number analyzed (Participants) | 23
  Peak viral load - Low < 1:40 | 4.7 [-1.5 to 14.8]
  Peak viral load - High >= 1:40: number analyzed (Participants) | 52
  Peak viral load - High >= 1:40 | 2.9 [-1.4 to 12.1]
  AUC - Low < 1:40: number analyzed (Participants) | 23
  AUC - Low < 1:40 | 4.6 [-2.2 to 14.8]
  AUC - High >= 1:40: number analyzed (Participants) | 52
  AUC - High >= 1:40 | 2.7 [-2.1 to 12.2]

39. Secondary Outcome: Percentage of Participants Reporting Any MMID Symptom During Challenge Period by Viral Shedding Status and Baseline HAI Seroprotection Status From Serum Measured at Baseline - RT-PCR Positive (One or More)
Description: Blood samples were collected pre-challenge (Day -2) for the HAI assay conducted with the A/Bethesda/MM2/H1N1 virus as the antigen. The geometric mean of each sample's replicate results was calculated from available results, then grouped by seroprotection status (titer results >= 1:40 vs < 1:40). The presence of any of the following symptoms was assessed from Day 2 to Day 8; body aches or pain, chest tightness, chills, conjunctivitis, nasal congestion, sinus congestion, coryza, decreased appetite, diarrhea, dry cough, dyspnea, fatigue, fever, headache, lymphopenia, nausea, a 3% or more decrease in oxygen saturation from baseline, productive cough, rhinorrhea, sore throat, and sweats. The percentage of participants that reported any symptom was calculated within each pre-challenge seroprotection status group and by viral shedding status, as observed anytime from Day 2 to Day 8; RT-PCR Negative (never positive), and at least once RT-PCR Positive.
Time Frame: Day 2 through Day 8
Population: All RT-PCR Positive (one or more) participants who received the study challenge, had a baseline sample for immunogenicity, and were followed for the entire duration of the study challenge period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 62
percentage of participants
  Any Symptom: Low < 1:40: number analyzed (Participants) | 36
  Any Symptom: Low < 1:40 | 83.3 [67.2 to 93.6]
  Any Symptom: High >= 1:40: number analyzed (Participants) | 26
  Any Symptom: High >= 1:40 | 92.3 [74.9 to 99.1]

40. Secondary Outcome: Percentage of Participants Reporting Any MMID Symptom During Challenge Period by Viral Shedding Status and Baseline HAI Seroprotection Status From Serum Measured at Baseline With RT-PCR Negative (None Positive)
Description: as for outcome 39
Time Frame: Day 2 through Day 8
Population: All RT-PCR Negative (none positive) participants who received the study challenge, had a baseline sample for immunogenicity, and were followed for the entire duration of the study challenge period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group
Number analyzed (Participants) | 14
percentage of participants
  Any Symptom: Low < 1:40: number analyzed (Participants) | 3
  Any Symptom: Low < 1:40 | 100 [29.2 to 100]
  Any Symptom: High >= 1:40: number analyzed (Participants) | 11
  Any Symptom: High >= 1:40 | 100 [71.5 to 100]

41. Secondary Outcome: Number of Serious Adverse Events (SAE) Post-challenge Through the Inpatient Stay
Description: SAEs included any untoward medical occurrence that resulted in death or a congenital anomaly/birth defect; was life threatening or a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation of existing hospitalization. All events are included regardless of relationship to the study challenge.
Time Frame: Day 1 through Day 8
Population: All participants who received the study challenge.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants | 0

42. Secondary Outcome: Number of Serious Adverse Events (SAE) Post- Inpatient Discharge Through the Duration of the Study
Description: SAEs included any untoward medical occurrence that resulted in death or a congenital anomaly/birth defect; was life threatening or a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation of existing hospitalization. All events are included regardless of relationship to the study challenge.This table provides the number and percentage of participants who reported SAEs following discharge from the study hospital.
Time Frame: Day 9 through Day 91
Population: All participants who received the study challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 76
Participants | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred from Receipt of Vaccination (Day 1) through final study visit (Day 91 +/- 7 days) were reported.
Description: Solicited AEs were assessed using MedDRA 22.0
Arm/Group | Group 1
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 41/76
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=76)
Lymphadenopathy (Blood and lymphatic system disorders) | 10 (10)
Tachycardia (Cardiac disorders) | 8 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5)
Alanine Aminotransferase Increased (Investigations) | 7 (11)
Blood Pressure Diastolic Decreased (Investigations) | 5 (8)
Blood Pressure Increased (Investigations) | 4 (4)
Blood Pressure Systolic Increased (Investigations) | 9 (15)
Platelet Count Increased (Investigations) | 7 (14)
Respiratory Rate Increased (Investigations) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT04044352/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT04044352/SAP_002.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT04044352/ICF_000.pdf